CLINICAL TRIAL: NCT01241019
Title: Safety and Efficacy of Oral Topiramate in Neonates With Hypoxic Ischemic Encephalopathy Treated With Hypothermia: a Pilot Study of the Neonatal Neuroprotection of Asphyxiated Tuscan Infants (NeoNATI) Network
Brief Title: Safety and Efficacy of Topiramate in Neonates With Hypoxic Ischemic Encephalopathy Treated With Hypothermia
Acronym: NeoNATI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Luca Filippi, Dr. Luca Filippi, Meyer Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT: 2010-018627-25
Record Dates: First submitted 2010-11-10; First posted 2010-11-16 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: asphyxia neonatorum, hypothermia, neuroprotection
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Asphyxia Neonatorum; Hypothermia | interventions — Topiramate; Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topiramate (Experimental): Newborns with hypoxic ischemic encephalopathy treated with mild hypothermia and topiramate
  Interventions: Drug: Topiramate in newborns with hypoxic ischemic encephalopathy treated with therapeutic hypothermia
- Control (No Intervention): Newborns with hypoxic ischemic encephalopathy treated with mild hypothermia

INTERVENTIONS:
Drug: Topiramate in newborns with hypoxic ischemic encephalopathy treated with therapeutic hypothermia — TPM 10 mg/kg once a day will be administered with an orogastric tube as enteric-coated granules mixed with water on arrival in the NICU, when the cooling will be begun (T0), once a day for the first 3 days of life, for a total of 3 doses per patient.
  Arms: Topiramate

SUMMARY:
The purpose of this study is to determine whether the administration of topiramate to newborns with hypoxic-ischemic encephalopathy potentiates the neuroprotective effect of treatment with hypothermia.

DETAILED DESCRIPTION:
Neonatal hypoxic-ischemic encephalopathy, due to perinatal asphyxia, is one of the leading causes of cerebral palsy, whose incidence, despite improvements in perinatal practice and neonatal care, has remained essentially unchanged over the recent past decades. It occurs approximately in 2-3 newborns every 1000 live births with a mortality rate of 10% for mild degrees and 60% for severe degrees. About 30% of survivors with mild hypoxic-ischemic encephalopathy and 100% with severe hypoxic-ischemic encephalopathy exhibit variable degrees of neurological disability.

Several studies have demonstrated the therapeutic effects of whole-body or selective head cooling to treat neonates with hypoxic-ischemic encephalopathy. Mild hypothermia, (rectal or esophageal temperature 33-34°C), started within 6 h after birth and protracted for 48-72 h, can significantly improve primary outcome measures such as death or disability at 18 months or improve the neurological outcome in survivors. Consequently, mild hypothermia is at present recommended for the treatment of moderate degrees of encephalopathy.

Topiramate an anticonvulsant agent widely used in adults and children, has been demonstrated to posses neuroprotective properties against hypoxic ischemic brain damage, both in vitro and in animal models and has been included in neuroprotective strategies for ischemic stroke and neonatal hypoxic-ischemic cerebral injury. Recently, topiramate treatment in asphyxiated newborns has been reported safe.

Aim of the present study is to confirm the safety and to evaluate whether the association of topiramate enhances the neuroprotective properties of hypothermia for the treatment of neonatal hypoxic-ischemic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age > 36 weeks and birth weigh > 1800 g with at least 1 of the following: a) Apgar score < 5 at 10 minutes; b) persisting need for resuscitation, including endotracheal intubation or mask ventilation 10 minutes after birth; c) acidosis (pH <7.0, base deficit >-16 mmol/L in umbilical cord blood or arterial, venous or capillary blood) within 60 minutes from birth;
2. moderate to severe encephalopathy, consisting of altered state of consciousness (irritability, lethargy, stupor, or coma) and > 1 of the following sings: a) hypotonia, b) abnormal reflexes, including oculomotor or pupil abnormalities, c) absent or weak suck, d) clinical seizures.
3. abnormal aEEG

Exclusion Criteria:

congenital abnormalities, congenital viral infections or evidence encephalopathy other than HIE.

-

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary aim is to evaluate the neurological outcome at 6, 12, 18 months of life | 18 months of life

SECONDARY OUTCOMES:
The secondary aim is to evaluate the efficacy of treatment with topiramate for improving neuroradiological outcome at 3 and 12 months of life | 12 months of life

CONTACTS AND LOCATIONS:
Overall Officials: Luca Filippi, MD, Principal Investigator — Azienda Ospedaliero-Universitaria A. Meyer, Firenze, Italy
Locations (2):
- Italy (2):
  - Neonatal Intensive Care Unit - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Neonatal Intensive Care Unit - Azienda Ospedaliero-Universitaria Pisana, Pisa

REFERENCES:
- [Background] Filippi L, la Marca G, Fiorini P, Poggi C, Cavallaro G, Malvagia S, Pellegrini-Giampietro DE, Guerrini R. Topiramate concentrations in neonates treated with prolonged whole body hypothermia for hypoxic ischemic encephalopathy. Epilepsia. 2009 Nov;50(11):2355-61. doi: 10.1111/j.1528-1167.2009.02302.x. Epub 2009 Sep 10. PMID 19744111
- [Background] Filippi L, Poggi C, la Marca G, Furlanetto S, Fiorini P, Cavallaro G, Plantulli A, Donzelli G, Guerrini R. Oral topiramate in neonates with hypoxic ischemic encephalopathy treated with hypothermia: a safety study. J Pediatr. 2010 Sep;157(3):361-6. doi: 10.1016/j.jpeds.2010.04.019. Epub 2010 May 31. PMID 20553846
- [Derived] Shankaran S. Outcomes of hypoxic-ischemic encephalopathy in neonates treated with hypothermia. Clin Perinatol. 2014 Mar;41(1):149-59. doi: 10.1016/j.clp.2013.10.008. PMID 24524452
- [Derived] Filippi L, Fiorini P, Daniotti M, Catarzi S, Savelli S, Fonda C, Bartalena L, Boldrini A, Giampietri M, Scaramuzzo R, Papoff P, Del Balzo F, Spalice A, la Marca G, Malvagia S, Della Bona ML, Donzelli G, Tinelli F, Cioni G, Pisano T, Falchi M, Guerrini R. Safety and efficacy of topiramate in neonates with hypoxic ischemic encephalopathy treated with hypothermia (NeoNATI). BMC Pediatr. 2012 Sep 5;12:144. doi: 10.1186/1471-2431-12-144. PMID 22950861
- See also: Drug information — http://druginfo.nlm.nih.gov/